CLINICAL TRIAL: NCT01176188
Title: A Nursing Intervention to Enhance Comfort and Promote Psychological Well-Being in Children During and Following PICU Hospitalization: A Pilot Study
Brief Title: A Nursing Intervention to Enhance Child Comfort and Psychological Well-Being During and Following PICU Hospitalization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Réseau de recherche portant sur les interventions en sciences infirmières du Québec (RRISIQ) (Unknown); Canadian Nurses Foundation (CNF) (Other)
Responsible Party: Principal Investigator, Dr. Janet Rennick, Nurse Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-069-PED
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Psychological Stress
Keywords: Pediatric Intensive Care Unit; Environmental Stressors; Sleep; Psychological Outcomes; Pediatrics
MeSH Terms: conditions — Stress, Psychological | interventions — Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comfort Care (Experimental): Parental soothing, including tactile and auditory strategies, followed by a quiet period with the application of earmuffs to block auditory stimulation
  Interventions: Other: Comfort Care
- Usual Care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Comfort Care — The intervention will consist of two parts: (1) A 15-20 minute period of parental soothing at the bedside comprised of calming activities which the child and parents are familiar with; (2) A quiet period will follow, in which earmuffs are applied over the child's ears to block auditory stimulation. The intervention will take place twice/24 hours, up to a maximum of 72 hours. Total time of first (daytime) intervention will be 2 hours, and of second (night-time) intervention will be 7 hours.
  Arms: Comfort Care
Other: Usual care — Usual nursing care for the child in the Pediatric Intensive Care Unit, including usual parental involvement and usual exposure to unit noise levels.
  Arms: Usual Care

SUMMARY:
Children who become critically ill and require Pediatric Intensive Care Unit (PICU)hospitalization may develop negative psychological outcomes following discharge. This pilot study will test a nursing intervention that seeks to promote child comfort, sleep and psychological well-being during and following PICU hospitalization.

Study objectives are to:

1. test the feasibility and acceptability of a PICU comfort care intervention that can be administered by nursing staff
2. examine the feasibility and acceptability of data collection procedures
3. pilot test outcome measures
4. determine effect sizes to inform sample size calculation for a future multi-centred randomized controlled trial (RCT).

The intervention will take place in the PICU, and consists of a parental soothing activity followed by a quiet period in which earmuffs are placed over the child's ears to block noise. Children's sleep time and comfort level will be monitored in the PICU, and the investigators will follow them for 3 months post-discharge to examine the effects of the intervention on psychological well-being.

DETAILED DESCRIPTION:
Background: Children who become critically ill and require Pediatric Intensive Care Unit (PICU) hospitalization may develop negative psychological outcomes following discharge. Despite this concern, there have been no systematic attempts to intervene with critically ill children to promote well-being, and prevent long term sequelae. The aim of this pilot study is to test the feasibility and acceptability of a PICU nursing intervention that seeks to enhance child comfort and promote sleep quality and duration in the PICU, potentially promoting psychological well-being post-discharge. The intervention is based on principles of Developmental Care, a philosophy of care that includes the child and family, and incorporates intervention strategies to reduce environmental stressors and improve quality of life. In view of the critically ill child's state of physical and emotional vulnerability, and the highly noxious environmental stimuli they are exposed to in the PICU, our proposed intervention has the potential to enhance physiological and psychological stability in this population. We will examine intervention effects on children's quality of sleep and sleep duration in the PICU, psychological distress post-PICU, and on parent anxiety during and following their child's PICU hospitalization.

Objectives: (1) To test the feasibility and acceptability of a PICU comfort care intervention that can be administered by nursing staff; (2) to examine the feasibility and acceptability of data collection procedures; (3) to pilot test outcome measures; and (4) to determine effect sizes to inform sample size calculation for a future multi-centred randomized controlled trial (RCT).

Design: A pilot study will be conducted using RCT design.

Outcomes: Results of this pilot study will provide essential information regarding feasibility of recruitment and randomization, as well as feasibility and acceptability of the developmental care intervention and data collection procedures - all of which will be incorporated into a full-scale RCT. While sample size is insufficient to allow statistical analyses, we will obtain initial estimates regarding changes in sleep duration, sleep fragmentation, and psychological well-being post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-17 admitted to the PICU of one Canadian, university teaching hospital
* Child in age-appropriate grade at school (+- 1 year)
* Child can read and speak English or French
* Parent or primary caregiver willing to participate in the intervention, who can read, speak and write English or French

Exclusion Criteria:

* Child diagnosed with a sleep disorder, seizure disorder, hearing disorder, or who has had neurological surgery that precludes sleep measurement
* Child expected to die during their PICU stay

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility of the comfort intervention | Time 1: Pediatric Intensive Care Unit, post-intervention: Time 2: Hospital Ward; Time 3: 3 months post-discharge

SECONDARY OUTCOMES:
Child Distress | 3 months post-Pediatric Intensive Care Unit discharge
Child Comfort | During Pediatric Intensive Care Unit stay
Parent Anxiety | Time 1: During child's Pediatric Intensive Care Unit stay; Time 2: 3 months post-discharge of child
Child Anxiety | 3 months post-discharge
Child Sleep | Time 1: During Pediatric Intensive Care Unit stay; Time 2: Hospital Ward; Time 3: 3 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Rennick, MSN, PhD, Principal Investigator — Montreal Children's Hospital, McGill University Health Center
Locations (1):
- Pediatric Intensive Care Unit, The Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Rennick JE, Stremler R, Horwood L, Aita M, Lavoie T, Majnemer A, Antonacci M, Knox A, Constantin E. A Pilot Randomized Controlled Trial of an Intervention to Promote Psychological Well-Being in Critically Ill Children: Soothing Through Touch, Reading, and Music. Pediatr Crit Care Med. 2018 Jul;19(7):e358-e366. doi: 10.1097/PCC.0000000000001556. PMID 29659416